CLINICAL TRIAL: NCT07219693
Title: QuantaFlo HD Clinical Validation Study
Status: Recruiting | Type: Observational
Sponsor: Semler Scientific (Industry)
Responsible Party: Sponsor
Other Study IDs: 35-0262-01
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: To Assess Cardiovascular Function
Keywords: cardiovascular function; transthoracic echocardiography; global longitudinal strain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: QuantaFlo HD — blood flow at the finger during a forced expiration

SUMMARY:
The primary aim of this validation protocol is to assess cardiovascular function through transthoracic echocardiography ("Echo") measurements and the QuantaFlo HD test measuring blood flow at the finger during a forced expiration ("FE"). The study examines whether Echo-measured GLS values greater than -16% correlate with abnormal responses during FE as measured by QuantaFlo HD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult (≥ age 22) subjects with a minimum of 1 of the following:
* A history of Cardiovascular Diseasei or PAD
* Recorded history of at least two of the following
* Hypertension
* Diabetes
* Hyperlipidemia

Exclusion Criteria:

* Unable to safely perform a forced expiration, or unable to obtain a technically adequate FE test result
* Subjects with a pacemaker or ICD with pacemaker function
* Terminal advanced illness
* Recent cardiothoracic surgery (within 12 months)
* Retinal eye disease with anticoagulants
* History of eye surgery, within 90 days
* Uncontrolled hypertension >180 mmHg systolic pressure or >100 mmHg diastolic pressure
* Subjects with severe tremors

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at three clinical sites: one primary care clinic and one cardiac clinic, both with established echo referral pathways, and one dedicated echo clinic.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity | From enrollment to the end of treatment is up to 1 week
  Evaluate the sensitivity and specificity of QuantaFlo HD test results to GLS findings.

SECONDARY OUTCOMES:
Accuracy | From enrollment to the end of treatment is up to 1 week
  Accuracy comparing QuantaFlo HD test results to GLS findings

CONTACTS AND LOCATIONS:
Locations (1):
- Pima Heart and Vascular, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No